CLINICAL TRIAL: NCT03177187
Title: ACE: Proof of Concept Phase I/II Trial of the CXCR2 Antagonist AZD5069, Administered in Combination with Enzalutamide, in Patients with Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Combination Study of AZD5069 and Enzalutamide.
Acronym: ACE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinuation of production of IMP
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Astellas Pharma Inc (Industry); AstraZeneca (Industry); Prostate Cancer UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR4500
Record Dates: First submitted 2017-05-26; First posted 2017-06-06 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide; enzalutamide

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I (Experimental): Increasing doses of AZD5069 in combination with a fixed dose of enzalutamide to establish the recommended phase II dose.
  Interventions: Drug: AZD5069; Drug: Enzalutamide 40 MG
- Phase II (Experimental): The Phase II part of the study will evaluate the recommended phase II dose identified in Phase I of the study in patients with metastatic castration resistant prostate cancer.
  RECRUITING
  Interventions: Drug: AZD5069; Drug: Enzalutamide 40 MG

INTERVENTIONS:
Drug: AZD5069 — 10mg and 40mg plain, beige, film-coated tablets packaged in bottles
Drug: Enzalutamide 40 MG — Enzalutamide is presented in 40mg white to off white capsules or tablets. The capsules/tablets are provided in a cardboard wallet incorporating a PVC/PCTFE/aluminium blister which holds 28 soft capsules/tablets. Each carton contains 4 wallets (112 soft capsules/tablets). Or tablets in bottles (120 per bottle).
  Other Names: Xtandi

SUMMARY:
ACE is a multi-centre proof of concept Phase I/II trial of the CXCR2 antagonist AZD5069, administered in combination with enzalutamide, in patients with metastatic castration resistant prostate cancer(mCRPC). The investigators will be investigating the safety and toxicity of the combination.

DETAILED DESCRIPTION:
The purpose of this study is to find out the side effects and safety of a combination of the CXCR2 antagonist, AZD5069 in combination with the androgen receptor antagonist, enzalutamide in patients with metastatic castration resistant prostate cancer and to determine the most appropriate dose of this combination. During the phase I study, patients will receive AZD5069 orally twice daily (BD) in combination with enzalutamide at 160mg orally once daily continuously. The starting dose of AZD5069 will be 40mg BD (dose level 1): other doses to be evaluated will include 80mg BD (dose level 2), 120mg BD (dose level 3), 160mg BD (dose level 4) and 320mg BD (dose level 5) in order to determine the MTD and RP2D to take forward to a Phase II reversal of resistance cohort. Intermediate dose levels such as 240mg BD may also be evaluated. During dose levels 1 to 4, patients will start with AZD5069 monotherapy for two weeks before commencing the combination. At all other dose levels, the two agents will be started concurrently. In addition, if agreed by the SRC, intermediate dose levels such as 240 mg taken BD will be explored. The Phase II part of the study will evaluate the optimized dose/schedule identified in Phase I of the study in patients with metastatic castration resistant prostate cancer.

In the Phase I part of the study, the AZD5069 is started first and will be taken twice daily as an oral tablet at Cycle 1, Day -14 for 14 days. Two weeks later on Cycle 1 Day 1, patients will start taking 160mg enzalutamide once a day in addition to the AZD5069. The starting dose of AZD5069 will be 40mg taken orally twice daily with single dose escalations to 80mg, 120mg and 160mg taken orally twice daily to determine the MTD to take forward to a Phase II reversal of resistance cohort.

The Phase II reversal of enzalutamide resistance study will explore whether the addition of AZD5069 to enzalutamide reverses resistance to enzalutamide alone. In the phase II reversal of enzalutamide resistance study patients will start taking the AZD5069 at the dose established in the Phase I safety run in part of the study in combination with 160mg of enzalutamide once a day and at the same time from Cycle 1 Day 1 onwards.

If the MTD of AZD5069 is greater than 160 mg BD, two different dose levels may be taken forward to the phase II study to determine efficacy. Only patients who have experienced disease progression after at least 12 weeks of treatment with enzalutamide, apalutamide or darolutamide will be eligible for this trial. Those patients who progressed on enzalutamide, apalutamide or darolutamide (at least 12 weeks of therapy) greater than 6 months prior to starting the IMP will enter the Phase II enzalutamide resistance run in cohort to confirm resistance to enzalutamide; once progression on enzalutamide is confirmed they will enter the Phase II reversal of enzalutamide resistance cohort.

Up to approximately 86 patients will be enrolled into this phase I/II trial, with up to 36 patients in the phase I safety run in cohort depending on number of patients required to determine the RP2D and up to 50 patients in the phase II study. We predict around 50% of these patients will enter the phase II enzalutamide resistance run in cohort first. The anticipated accrual rate for this trial is 3-6 patients per month across 4 centres.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and be capable of cooperating with treatment.
2. Age ≥ 18 years
3. Histologically confirmed adenocarcinoma of the prostate and with tumour tissue accessible for research analysis for this trial. Patients who have no histological diagnosis must be willing to undergo a biopsy to prove prostate adenocarcinoma.
4. Metastatic castration resistant prostate cancer.
5. Documented prostate cancer progression as assessed by the investigator with RECIST (v1.1) and PCWG2 criteria (section 3.6) with at least one of the following criteria:

   a. Progression of soft tissue/visceral disease by RECIST (v1.1) and/or, b. Progression of bone disease by PCWG2 bone scan criteria and/or, c. Progression of PSA by PCWG2 PSA criteria and/or, d. Clinical progression with worsening pain and need for palliative radiotherapy for bone metastases.
6. PSA ≥ 10ng/ml.
7. Received prior castration by orchiectomy and/or ongoing luteinizing hormone releasing hormone agonist treatment.
8. Ongoing androgen deprivation with serum testosterone < 50 ng/dL (<2.0 nM).
9. Willing to have pre- and post-treatment biopsies to obtain proof of mechanism from translational studies. Archival tissue must be available for research analysis
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
11. Documented willingness to use an effective means of contraception while participating in the study and for 6 months post last treatment dose as defined in section 9.6.
12. Able to swallow the study drug.
13. All efforts should be made to discontinue steroid usage but up-to 5mg BD prednisolone (or equivalent) will be allowed.
14. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.

    Laboratory Test Value required Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L WBC ≥ 3.0 x 109/L Calculated creatinine clearance ≥ 50 mL/min (uncorrected value) Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) unless documented Gilbert's disease. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)

    ≤ 2.5 x (ULN) unless raised due to known metastatic liver disease in which case ≤ 5 x ULN is permissible
15. Phase I safety run in cohort ONLY Patients that have progressed after either enzalutamide, apalutamide, darolutamide or abiraterone treatment (having received a minimum of 12 weeks of enzalutamide, apalutamide, darolutamide or abiraterone treatment).
16. Patients with histologically confirmed adenocarcinoma of the prostate that have progressed after either enzalutamide, apalutamide or darolutamide (having received a minimum of 12 weeks of enzalutamide, apalutamide or darolutamide) more than 6 months prior to entry (day of starting IMP). Prior treatment with abiraterone is not an exclusion criteria.
17. Patients with histologically confirmed adenocarcinoma of the prostate that have progressed after either enzalutamide. apalutamide or darolutamide (having received a minimum of 12 weeks enzalutamide, apalutamide or darolutamide ) within 6 months prior to entry (day of starting IMP). Prior treatment with abiraterone is not an exclusion criteria.

Exclusion Criteria:

* 1. Surgery, chemotherapy or other anti-cancer therapy within 4 weeks prior to trial entry/randomization into the study (with the exception of enzalutamide, apalutamide or darolutamide). Any other therapy for prostate cancer, other than gonadotropin releasing hormone analogue therapy, such as progesterone, medroxyprogesterone, progestins or 5-alpha reductase inhibitors, must be discontinued at least 2 weeks before the first dose of the study drug.

  2. Participation in another interventional clinical trial of an IMP within 4 weeks prior to trial entry. Participation in trials of licenced medications is allowed provided the medication is not a prohibited concomitant medication.

  3. Prior limited field radiotherapy within 2 weeks and wide field radiotherapy within 4 weeks prior to trial entry.

  4. Clinical and/or biochemical evidence of hyperaldosteronism or hypopituitarism.

  5. History of seizures or other predisposing factors including, but not limited to, underlying brain injury, stroke, primary brain tumours, brain metastases and leptomeningeal disease, or alcoholism.

  6. Use of potent inhibitors/inducers of CYP3A4, CYP2C9 and CYP2C19 should be avoided during the trial and 4 weeks prior to trial entry.

Co-administration of drugs that are known potent or moderate CYP3A4 inhibitors, potent or moderate CYP3A4 inducers (with the exception of enzalutamide), P-gp substrates with narrow therapeutic index, sensitive CYP2B6 substrates, warfarin or any other coumarin derivative, BCRP-substrates that reduce blood neutrophils, Seville orange or grapefruit products.

Use of herbal medications during the trial and 4 weeks afterwards. 7. Malabsorbtion syndrome or other condition that would interfere with enteral absorption.

8. Any of the following cardiac criteria:

* • QT interval > 470 msec.
* Clinically important abnormalities including rhythm, conduction or ECG changes (left bundle branch block, third degree heart block).
* Factors predisposing to QT prolongation including heart failure, hypokalemia, congenital long QT syndrome, family history of prolonged QT syndrome, unexplained sudden death (under 40) and concomitant medications known to prolong QT interval.
* Coronary artery bypass, angioplasty, vascular stent, myocardial infarction, angina or congestive heart failure (NYHA ≥ grade 2) in the last 6 months (see appendix 4 for NYHA scale).
* Uncontrolled hypotension (systolic blood pressure < 90mmHg and or diastolic blood pressure < 50 mmHg).
* Uncontrolled hypertension on optimal medical management 9. Clinically significant history of liver disease (Chlid-Pugh B or C, viral or other hepatitis, current alcohol abuse or cirrhosis).

  10. Any other finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect interpretation of the results or renders the patients at high risk from treatment complications e.g patients with a hypersensitivity to the active substance or any of the excipients.

  11. Malignancy other than prostate cancer within 5 years of trial entry with the exception of adequately treated basal cell carcinoma.

  12. Unresolved significant toxicity from prior therapy (except alopecia and grade 1 peripheral neuropathy).

  13. Inability to comply with study and follow-up procedures. 14. Patients with predominantly small cell or neuroendocrine differentiated prostate cancer are not eligible.

  15. Immunocompromised patients. 16. Active or uncontrolled autoimmune disease requiring corticosteroid therapy.

  17. History of thromboembolic disease within 12 months of commencement of trial.

  18. At high-risk because of non-malignant systemic disease including active infection and any serious concurrent illness.

  19. Any known intolerance to enzalutamide, AZD5069 or to any constituents

  20. Symptoms of COVID-19 and/or documented COVID-19 infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 30 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) in Phase I of AZD5069 administered in combination with enzalutamide at 160mg OD. | 12 months
  The maximum dose at which no more than 1 of 6 patients at same dose level experience a drug related toxicity (DLT), as defined in the protocol.
Antitumour activity of AZD5069 in combination with enzalutamide as measured by response rate in Phase II | 12 months
  * Prostate specific antigen (PSA) decline ≥ 50% criteria confirmed 4 weeks or later and/or,
  * Confirmed soft tissue objective response by RECIST (v1.1) in patients with measurable disease and/or,
  * ONLY for patients with detectable circulating tumour cell count (CTC) of ≥ 5/7.5ml blood at baseline, conversion of CTC <5/7.5ml blood nadir.
Antitumour activity of AZD5069 in combination with enzalutamide as measured by response rate in Phase II | 12 months
  For disease progression (see section 3.6) the Prostate Cancer Working Group 2 (PCWG2) criteria and RECIST (v1.1) criteria will be used. Treatment failure will be defined as:
  * Progression of soft tissue/visceral disease by RECIST (v1.1) and/or,
  * Progression of bone disease by PCWG2 bone scan criteria and/or
  * Progression of PSA by PCWG2 PSA criteria.

SECONDARY OUTCOMES:
PSA decline | 24 months
  Maximal PSA decline at any time during the trial and PSA decline after 12 weeks (as per PCWG2 criteria) of combination treatment.
Overall survival of patients in Phase II | 24 months
  Overall survival will be measured from the date of AZD5069 addition to enzalutamide to the date of death (whatever cause). Survival time of living patients will be censored on the last date of patient is known to be alive or lost to follow up.
To estimate the radiologic progression free survival (rPFS) on the combination in Phase II | 24 months
  rPFS will be measured from the date of AZD5069 addition to enzalutamide until:
  * Progression of soft tissue/visceral disease by RESIST and/or,
  * Progression of bone disease by PCWG2 bone scan criteria and/or,
  * Death of any cause
  Patients withdrawn for any reason prior to radiological progression then the patient should be assessed until radiological progression has occurred. If however they have started another treatment then they will be censored at the start of the new treatment.
To assess the effects of AZD5069 and enzalutamide on the number of circulating tumour cells in Phase II | 24 months
  CTC fall by >30% will be expressed as the proportion of patients that have demonstrated a CTC fall of >30% after 12 weeks of combination treatment.
To further evaluate the safety and tolerability of the combination in patients who progress on enzalutamide in Phase II | 24 months
  Recording the population exposure to the AZD5069 and enzalutamide combination will summarise safety. Adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
To further characterise the PD profile of AZD5069 and enzalutamide when administered in combination in Phase II | 24 months
  Number of patients with a neutrophil to lymphocyte ratio (NLR) ≥ 3 (at baseline) that convert to an NLR < 3 (blood nadir) with AZD5069 and enzalutamide in combination.
To characterise the pharmacokinetic (PK) profile of enzalutamide and AZD5069 when administered in combination in Phase I | 24 months
  Plasma concentration of enzalutamide and AZD5069 in whole blood
To characterise the pharmacodynamic (PD) profile of AZD5069 and enzalutamide when administered in combination in Phase I | 24 months
  Number of patients with a neutrophil to lymphocyte ratio (NLR) ≥ 3 (at baseline) that convert to an NLR < 3 (blood nadir) with AZD5069 and enzalutamide in combination.
To estimate the antitumour activity of AZD5069 in combination with enzalutamide as measured by response rate in Phase I. | 24 months
  Antitumour activity will be defined by response rate on the basis of the following outcomes; if any of these occur, patients will be considered to have responded:
  * PSA decline ≥ 50% criteria confirmed 4 weeks or later and/or,
  * Confirmed soft tissue objective response by RECIST (v1.1) in patients with measurable disease and/or,
  * ONLY for patients with detectable circulating tumour cell count (CTC) of ≥ 5/7.5ml blood at baseline, conversion of CTC <5/7.5ml blood nadir.
To further characterise the PD profile of AZD5069 and enzalutamide when administered in combination in Phase II | 24 months
  Number of patients patients whose circulating myeloid derived suppressor cells (MDSCs) and intratumoral MDSCs reduce by 50% with AZD5069 and enzalutamide in combination.
To characterise the pharmacodynamic (PD) profile of AZD5069 and enzalutamide when administered in combination in Phase I | 24 months
  Number of patients whose circulating myeloid derived suppressor cells (MDSCs) and intratumoral MDSCs reduce by 50% with AZD5069 and enzalutamide in combination.
To estimate the antitumour activity of AZD5069 in combination with enzalutamide as measured by response rate in Phase I. | 24 months
  For disease progression (see section 3.6) the PCWG2 criteria and RECIST (v1.1) criteria will be used. Treatment failure will be defined as:
  * Progression of soft tissue/visceral disease by RECIST (v1.1) and/or,
  * Progression of bone disease by PCWG2 bone scan criteria and/or
  * Progression of PSA by PCWG2 PSA criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Johann De Bono, MD, Principal Investigator — National Health Service, United Kingdom
Locations (4):
- Bellinzona Hospital, Bellinzona, Switzerland
- United Kingdom (3):
  - Belfast City Hospital, Belfast, UK
  - The Royal Marsden Hospital Foundation Trust, Sutton, UK
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo C, Sharp A, Gurel B, Crespo M, Figueiredo I, Jain S, Vogl U, Rekowski J, Rouhifard M, Gallagher L, Yuan W, Carreira S, Chandran K, Paschalis A, Colombo I, Stathis A, Bertan C, Seed G, Goodall J, Raynaud F, Ruddle R, Swales KE, Malia J, Bogdan D, Tiu C, Caldwell R, Aversa C, Ferreira A, Neeb A, Tunariu N, Westaby D, Carmichael J, Fenor de la Maza MD, Yap C, Matthews R, Badham H, Prout T, Turner A, Parmar M, Tovey H, Riisnaes R, Flohr P, Gil J, Waugh D, Decordova S, Schlag A, Cali B, Alimonti A, de Bono JS. Targeting myeloid chemotaxis to reverse prostate cancer therapy resistance. Nature. 2023 Nov;623(7989):1053-1061. doi: 10.1038/s41586-023-06696-z. Epub 2023 Oct 16. PMID 37844613